CLINICAL TRIAL: NCT07018271
Title: A Study on the Use of Sulpegfilgrastim to Prevent the Incidence of Neutropenia With Infection in Newly Diagnosed Non-transplant Multiple Myeloma Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sulpegfilgrastim in NDMM
Record Dates: First submitted 2025-05-27; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; DRD; Sulpegfilgrastim; Neutropenia
MeSH Terms: conditions — Multiple Myeloma; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): On Day 1 of each oncological treatment cycle, after administration of the CD38 monoclonal antibody, a subcutaneous injection of Sulfubrolipoyl G-CSF will be given. The recommended fixed dose of Sulfubrolipoyl G-CSF is 6 mg per injection. The study will observe six treatment cycles. After the study concludes, the next treatment steps will be jointly decided by the investigator and the patient.
  Interventions: Drug: sulpegfilgrastim

INTERVENTIONS:
Drug: sulpegfilgrastim — On Day 1 of each oncological treatment cycle, after administration of the CD38 monoclonal antibody, a subcutaneous injection of Sulfubrolipoyl G-CSF will be given. The recommended fixed dose of Sulfubrolipoyl G-CSF is 6 mg per injection.

SUMMARY:
The goal of this study is to observe and evaluate the incidence of infection in newly diagnosed, non-transplanted multiple myeloma patients receiving prophylactic treatment with sulpegfilgrastim (a pegylated recombinant human granulocyte colony-stimulating factor).

DETAILED DESCRIPTION:
It is a study on the use of sulpegfilgrastim to prevent the incidence of neutropenia with infection in newly diagnosed non-transplant multiple myeloma patients. Patients enrolled in this study may be treated with the following oncological protocols:DRD regimen (CD38 monoclonal antibody + lenalidomide + dexamethasone).On Day 1 of each oncological treatment cycle, after administration of the CD38 monoclonal antibody, a subcutaneous injection of Sulfubrolipoyl G-CSF will be given. The recommended fixed dose of Sulfubrolipoyl G-CSF is 6 mg per injection. The study will observe six treatment cycles. After the study concludes, the next treatment steps will be jointly decided by the investigator and the patient. If a patient's neutrophil level remains below 0.5×10⁹/L for over 24 hours after receiving Sulfubrolipoyl G-CSF, the investigator will assess the need for rescue treatment with short-acting G-CSF based on the patient's condition until the neutrophil level returns to normal.Prophylactic antibiotic treatment may be administered before the onset of oncological treatment. The goal is to observe and evaluate the incidence of infection in newly diagnosed, non-transplanted multiple myeloma patients receiving prophylactic treatment with sulpegfilgrastim (a pegylated recombinant human granulocyte colony-stimulating factor).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible for this study:

1. Age ≥ 18 years old，weight > 35 kg，regardless of gender;
2. Voluntarily participating in the study after signing the informed consent form;
3. Newly diagnosed, non-transplanted multiple myeloma patients diagnosed according to the 2016 International Myeloma Working Group (IMWG) criteria or the 2024 Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma, and expected to receive at least six cycles of DRD (CD38 monoclonal antibody + lenalidomide + dexamethasone) oncological treatment;
4. Deemed suitable for sulpegfilgrastim administration by the investigator;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2, with an expected survival of at least three months;
6. Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; platelet count (PLT) ≥ 75.0×10⁹/L；
7. Serum creatinine clearance rate ≥30 mL/min; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤three times the upper limit of normal。
8. Negative pregnancy test for women of childbearing age. Patients and their spouses must agree to use effective contraceptive measures during treatment and for one year thereafter；
9. Signed informed consent for chemotherapy. In cases where the patient is unable to sign due to impaired consciousness, upper limb paralysis, or illiteracy, a legal representative may sign on their behalf.

Exclusion Criteria:

Patients meeting any of the following criteria are excluded from this study：

1. Weight≤35kg；
2. Monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma, or primary light chain amyloidosis with organ involvement;
3. Diagnosed or treated for another malignancy within one year prior to registration, or evidence of residual disease from a previous malignancy requiring ongoing treatment;
4. Known positive for human immunodeficiency virus (HIV);
5. Pregnant or breastfeeding women;
6. Patients with any active acute infection, including viral infections;
7. Patients who have received systemic antibiotic treatment within two weeks prior to enrollment;
8. Allergy to Sulfubrolipoyl G-CSF, pegylated recombinant human granulocyte colony-stimulating factor, recombinant human granulocyte colony-stimulating factor, or other agents expressed in E. coli; Other situations where the investigator deems participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection during oncological treatment | through study completion, an average of 6 months
  Incidence of infection during oncological treatment

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) | through study completion, an average of 6 months
  Incidence of febrile neutropenia (FN)
Incidence of infection in patients with ANC <1.0×10⁹/L | through study completion, an average of 6 months
  Incidence of infection in patients with ANC <1.0×10⁹/L
Proportion of patients requiring dose adjustment due to ANC reduction or infection | through study completion, an average of 6 months
  Proportion of patients requiring dose adjustment due to ANC reduction or infection
Incidence of Grade 3 or higher ANC reduction in the first treatment cycle | through study completion, an average of 6 months
  Incidence of Grade 3 or higher ANC reduction in the first treatment cycle
Incidence of Grade 3 or higher ANC reduction across all observation cycles | through study completion, an average of 6 months
  Incidence of Grade 3 or higher ANC reduction across all observation cycles
Proportion of patients experiencing treatment delays (≥7 days) due to infection or neutropenia | through study completion, an average of 6 months
  Proportion of patients experiencing treatment delays (≥7 days) due to infection or neutropenia
Clinical efficacy of treatment in patients, VGPR rate, CR rate, MRD negative rate | through study completion, an average of 6 months
  Clinical efficacy of treatment in patients, VGPR rate, CR rate, MRD negative rate
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

IPD SHARING:
Plan to Share IPD: Yes
To observe and evaluate the incidence of infection in newly diagnosed, non-transplanted multiple myeloma patients receiving prophylactic treatment with sulpegfilgrastim (a pegylated recombinant human granulocyte colony-stimulating factor).
Supporting Information: Study Protocol